CLINICAL TRIAL: NCT02509143
Title: High-dose Acupuncture for Prevention of Postoperative Nausea and Vomiting in Patients Undergoing Laparoscopic Colorectal Surgery: A Randomized Controlled Pilot Study
Brief Title: Acupuncture for Postoperative Nausea and Vomiting in Patients Undergoing Colorectal Surgery
Acronym: AcuPONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Collaborators: Korea Institute of Oriental Medicine (Other Government); Korean Medicine Hospital of Pusan National University (Other)
Responsible Party: Principal Investigator, Kim Hee Young, Assistant Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 03-2015-010
Record Dates: First submitted 2015-07-17; First posted 2015-07-27 (Estimated); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Postoperative Nausea and Vomiting; Colorectal Neoplasms
Keywords: Postoperative Nausea and Vomiting; Colorectal Neoplasms
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Colorectal Neoplasms | interventions — Acupuncture Therapy; Antiemetics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High-dose acupuncture with intravenous infusion of ramosetron (Experimental): Three sessions of acupuncture on the points of Stomach 36 (ST36), Stomach 37 (ST37), Liver 3 (LR3), Large Intestine 11 (LI11), Large Intestine 4 (LI4), Spleen 6 (SP6), Spleen 4 (SP4), Pericardium 6 (PC6), Heart 8 (HT8), and Gall Bladder 41 (GB41) within 48 hours after surgery
  Interventions: Procedure: High-dose acupuncture with intravenous infusion of ramosetron; Device: P6 stimulation with intravenous infusion of ramosetron; Drug: Intravenous infusion of ramosetron
- P6 stimulation with intravenous infusion of ramosetron (Active Comparator): P6 stimulation by wearing a study wristband within 48 hours after surgery
  Interventions: Device: P6 stimulation with intravenous infusion of ramosetron; Drug: Intravenous infusion of ramosetron
- Intravenous infusion of ramosetron (Active Comparator): A mixture of standard antiemetic medication (5-Hydroxytryptophan receptor antagonist; ramosetron hydrochloride 0.3 mg) and analgesics, including anon-steroidal anti-inflammatory drug (NSAID) (ketorolac tromethamine 120 mg), and a semi-synthesized opioid (oxycodone 20 mg), will be infused by intravenous patient-controlled analgesia (1ml bolus/20 min lockout, 1ml/hr continuous infusion).
  Interventions: Drug: Intravenous infusion of ramosetron

INTERVENTIONS:
Procedure: High-dose acupuncture with intravenous infusion of ramosetron — Three sessions of acupuncture will be provided within 48 hours after surgery. Electrical stimulation with an alternating frequency of 2 to 100 Hz will be applied to selected points (PC6 to LI4, ST36 to ST37, and bilateral SP6).
  An embedded acupuncture technique for preoperative anxiety will be applied to the bilateral acupuncture points of Liver (LI4), Heart 7 (HT7), Stomach (ST36), Yin-Tang, ear Shen-Men,and ear sympathetic and will be removed the next day. Treatments will be provided by qualified hospital staff (Korean medical doctors) with more than 10 years of clinical experience. The same stimulation of P6 points and antiemetics will be provided to the P6 acupuncture-point stimulation group.
  Other Names: Acupuncture
  Arms: High-dose acupuncture with intravenous infusion of ramosetron
Device: P6 stimulation with intravenous infusion of ramosetron — Stimulation of P6 points will be maintained from one hour before and for 48 hours after surgery by wearing a wristband that produces pulse-type transcutaneous electrical stimulation. Antiemetics will be provided, the same as the standard antiemetic medication alone group.
  Other Names: PC6
  Arms: High-dose acupuncture with intravenous infusion of ramosetron; P6 stimulation with intravenous infusion of ramosetron
Drug: Intravenous infusion of ramosetron — Intravenous infusion of (oxycodone 20mg, ketorolac 120mg, ramosetron 0.3mg) as standard antiemetic medication will be provided. A dose of continuous infusion will be reduced by 0.1 ml/hr when a patient complaints of nausea.
  When vomiting occurs, a dose of continuous infusion will be reduced by 0.2 ml/hr and a bolus infusion of ramosetron 0.3 mg will be provided. A bolus infusion of ramosetron 0.3 mg will be also given if a patient feels greater than or equal to six points of nausea as measured on a 0 to 10 numeric rating scale (NRS) (nausea-severity scale) or by the patient's request, regardless of the severity of the nausea.
  Other Names: Antiemetics

SUMMARY:
Background: PONV is one of the prevalent discomforts in the early phase of recovery after surgery. Evidence suggests that the stimulation of the P6 acupuncture point can reduce the occurrence of PONV. What remains unclear is whether a higher dose of acupuncture produces more benefits compared with P6 stimulation alone or whether acupuncture combined with standard antiemetic medication yields better outcomes.

Objectives: This study aims to assess the effectiveness, safety, and feasibility of intensive acupuncture treatments combined with standard antiemetic medication as compared with P6 acupoint stimulation combined with standard antiemetic medication or with standard antiemetic medication alone.

DETAILED DESCRIPTION:
Background: PONV is one of the prevalent discomforts in the early phase of recovery after surgery. Evidence suggests that the stimulation of the P6 acupuncture point can reduce the occurrence of PONV. What remains unclear is whether a higher dose of acupuncture produces more benefits compared with P6 stimulation alone or whether acupuncture combined with standard antiemetic medication yields better outcomes. This study aims to assess the effectiveness and safety of different acupuncture regimen for the prevention of PONV: high-dose acupuncture treatments combined with standard antiemetic medication, P6 acupuncture-point stimulation combined with standard antiemetic medication, or medication alone.

Objectives: This study aims to assess the effectiveness, safety, and feasibility of intensive acupuncture treatments combined with standard antiemetic medication as compared with P6 acupoint stimulation combined with standard antiemetic medication or with standard antiemetic medication alone, to prevent postoperative nausea and vomiting (PONV) in patients undergoing laparoscopic colorectal surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective laparoscopic surgery of colorectal cancer resection (right hemicolectomy, left hemicolectomy, anterior resection with primary anastomosis, and low anterior resection with loop ileostomy for fecal diversion)
* Patients aged 18 to 80
* American Society of Anesthesiologists Grade 1 to 2
* Written informed consents

Exclusion Criteria:

* Pregnancy
* Inflammatory bowel disease
* Comorbidities that may affect outcomes of surgery (e.g., chronic kidney disease, chronic liver disease, cardiopulmonary failure, and diabetes with complications)
* Use of emetogenic / antiemetic medication within 24 hours before surgery
* Previous history of emetic episodes after administration of antibiotics
* Expected use of mechanical ventilation
* Cognitive impairment that may affect the patient's ability to complete the outcome assessments
* Previous history of stroke
* Previous history of sensitive reaction to acupuncture
* Patients unable to cooperate with acupuncture treatments
* Pacemaker implantation
* Previous history of epilepsy
* Patients who have received Korean medicine treatments (acupuncture, moxibustion, cupping, or herbal medicine) within 2 weeks
* Patients who have participated in other trials within 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Number of patients who experience moderate or severe level nausea or vomiting | at 24 hours after surgery
  Number of patients who experience moderate or severe level nausea (i.e, at least 4 points of nausea on 0 to 10 numeric rating scale) or vomiting during the first 24 postoperative hours

SECONDARY OUTCOMES:
Nausea scores on a numeric rating scale | at baseline (the discharge of recovery room), 6, 12, 24, 48 hours from baseline and at discharge (until discharge, an expected average of 7 days after surgery)
  Score ranges from 0 (no nausea at all) to 10 (the worst nausea imaginable)
Number of vomiting | from the discharge of recovery room to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 48 hours, 48 hours to the discharge (until discharge, an expected average of 7 days after surgery)
  Number of vomiting
Cumulative incidence of vomiting | at baseline to 24 and 48 hours
  Cumulative incidence of vomiting
Number of patients who experience nausea | from the discharge of recovery room to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 48 hours, 48 hours to the discharge (until discharge, an expected average of 7 days after surgery)
  Number of patients who experience nausea
Cumulative number of patients who experience nausea | at baseline to 24 and 48 hours
  Cumulative number of patients who experience nausea
Number of patients who experience vomiting | from the discharge of recovery room to 6 hours, 6 to 12 hours, 12 to 24 hours, 24 to 48 hours, 48 hours to the discharge (until discharge, an expected average of 7 days after surgery)
  Number of patients who experience vomiting
Cumulative number of patients who experience vomiting | at baseline to 24 and 48 hours
  Cumulative number of patients who experience vomiting
Pain scores on a numeric rating scale | at 6, 12, 24, 48 hours from the discharge of recovery room and at discharge (until discharge, an expected average of 7 days after surgery)
  Score ranges from 0 (no nausea at all) to 10 (the worst nausea imaginable)
Patient's global assessment of recovery after surgery | at 2 weeks after surgery
  Response options include very much improved, somewhat improved, no change, somewhat worsened, and very much worsened.
Time to first flatus | until discharge, an expected average of 7 days after surgery
  Time to first flatus
Time to tolerate soft diet | until discharge, an expected average of 7 days after surgery
  Time to tolerate soft diet
Time to first defecation | until discharge, an expected average of 7 days after surgery
  Time to first defecation
Time to independent walk | until discharge, an expected average of 7 days after surgery
  Time to independent walk
Number of insertions of nasogastric tube | until discharge, an expected average of 7 days after surgery
  Number of insertions of nasogastric tube
Time to first removal of Foley catheter | until discharge, an expected average of 7 days after surgery
  Time to first removal of Foley catheter
Number of reinsertions of Foley catheter | until discharge, an expected average of 7 days after surgery
  Number of reinsertions of Foley catheter
Number of clean intermittent catheterizations | until discharge, an expected average of 7 days after surgery
  Number of clean intermittent catheterizations
Quality of life measured by European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ) C30 | at 2 weeks after surgery
  Quality of life measured by European Organization for Research and Treatment
Preoperative anxiety | just before the induction of anaesthesia
  measured by 0 to 10 numeric rating scale (0: no anxiety, 10: extreme anxiety)
Patient-reported satisfaction for management of PONV | at 48 hours after surgery
  measured by 0 to 10 numeric rating scale (0: very unsatisfactory, 10: very satisfactory)
Use of medication | at 2 weeks after surgery
  Use of medication
Postoperative complications | within 4 weeks after surgery
  * wound infection
  * urinary tract infection
  * urinary retention
  * chest infection
  * other infection
  * paralytic ileus
Serious adverse events | within 4 weeks after surgery
  * respiratory failure requiring ventilation
  * renal failure requiring dialysis
  * cardiac failure
  * myocardial infarction
  * anastomotic leakage requiring surgery
  * anastomotic leakage requiring drainage
  * bowel obstruction/stricture requiring surgery
  * abdominal wall dehiscence requiring surgery
  * readmission within 30 days after surgery
  * reoperation within 30 days after surgery
  * mortality during surgery or within 30 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Hee Young Kim, PhD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (2):
- South Korea (2):
  - National Clinical Research Center, Korean Medicine Hospital, Pusan National University, Yangsan, Kyung Sang South Province
  - Pusan National University Yangsan Hospital, Yangsan, Kyung Sang South Province

REFERENCES:
- [Derived] Kim KH, Kim DH, Bae JM, Son GM, Kim KH, Hong SP, Yang GY, Kim HY. Acupuncture and PC6 stimulation for the prevention of postoperative nausea and vomiting in patients undergoing elective laparoscopic resection of colorectal cancer: a study protocol for a three-arm randomised pilot trial. BMJ Open. 2017 Jan 4;7(1):e013457. doi: 10.1136/bmjopen-2016-013457. PMID 28052910